CLINICAL TRIAL: NCT07306728
Title: Effect of Femoral Region Ice Bag Application on Patients' Clinical Outcomes
Brief Title: Effect of Femoral Region Ice Bag Application on Patients' Clinical Outcomes Post-Percutaneous Coronary Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hussein Abdeltawab Abdelmoneim Hussein Glalah, Nursing specialist, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29806151204272
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease(CAD); Percutaneous Coronary Intervention
Keywords: Ice Bag Application, Clinical Outcomes, Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice Bag Application (IBA) Group (Other): Patients in this group will receive localized cold therapy, consisting of an ice bag maintained at a temperature of 0-4°C, applied to the femoral region for 20 minutes with 10-minute intervals during the first two hours following PCI
  Interventions: Other: Ice Bag Application
- • Routine Care Group (No Intervention): Patients in this group will receive standard post-PCI care as per hospital protocol, which includes the application of a sandbag to the femoral site for 20 minutes with 10-minute intervals during the first two hours following PCI.

INTERVENTIONS:
Other: Ice Bag Application — cold therapy, consisting of an ice bag maintained at a temperature of 0-4°C, applied to the femoral region for 20 minutes with 10-minute intervals during the first two hours following PCI
  Arms: Ice Bag Application (IBA) Group

SUMMARY:
Coronary artery disease (CAD) remains a leading cause of morbidity and mortality worldwide, necessitating advancements in diagnostic techniques (Parulkar et al., 2025). According to the British Heart Foundation, over 250 million individuals worldwide are living with CAD, making it the most commonly diagnosed heart condition globally. In 2021, CAD was responsible for approximately 9 million deaths, accounting for about one in every seven deaths globally

DETAILED DESCRIPTION:
Complications associated with PCI significantly impact patient outcomes and place substantial demands on healthcare systems. These adverse events contribute to increased morbidity and mortality rates, prolonged hospitalizations, higher healthcare expenditures, and longer 0waiting times for subsequent cardiac procedures. (Guedeney et al., 2024; Ntow, Agyeman, Aryal, & Patel, 2024) . Postoperative pain remains a prevalent concern following PCI, particularly after femoral catheter removal, with approximately 33% of patients reporting discomfort at the access site (Al-Zuhairi & Abed, 2024).

Although this pain typically subsides over time, it can significantly affect patient comfort and recovery in the immediate post-procedural phase. In addition to pain, hematoma formation is among the most frequent vascular complications associated with femoral artery access, with a reported prevalence of up to 15.5% (Zhi et al., 2024). These hematomas, resulting from bleeding at the puncture site, can range from minor bruising to substantial blood collections, potentially leading to pain, swelling, and further clinical complications (Hamdi, Abd El Megeed, Abd Al Ghaffare, & Abdelmowla, 2023). Traditional pressure application remains a commonly employed strategy in clinical settings for managing such hematomas and mitigating their progression (Rodgers et al., 2025).

Cryotherapy, or cold therapy, is a well-established non-pharmacological intervention widely utilized in clinical practice to alleviate pain, reduce swelling, and control inflammation. This method typically involves the localized application of ice packs or bags, which may range from specially designed medical devices to simple waterproof plastic bags (Garcia, Karri, Zacharias, & Abd-Elsayed, 2021). In the context of PCI care, cryotherapy has shown promise in minimizing vascular complications following femoral arterial sheath removal. The application of a cold pack to the femoral region can aid in reducing pain, controlling bleeding, and limiting hematoma formation.

The therapeutic effect is primarily attributed to the vasoconstriction induced by cold exposure, which enhances coagulation, decreases local blood flow, and increases blood viscosity (Al-Bayati & Al-Kassar, 2023). Additionally, it decreases temperature by primarily reducing metabolic activity, which reduces inflammatory response as well as reduces nerve conductivity, thereby slowing pain impulse transmission and decreasing pain perception and tissue damage (Behera & Shetty, 2023).

The significance of this study lies in its potential to enhance post-PCI patient care through a simple, non-pharmacological intervention. Growing evidence supports the clinical effectiveness of ice bag application in managing complications associated with femoral catheter removal. Research by )Al-Zuhairi and Abed 2024), and )Pamuk and Özkaraman 2024), confirmed that localized ice therapy significantly alleviates pain and reduces vascular complications following PCI, emphasizing its role in improving patient comfort and outcomes.

Furthermore, findings by (Suhanda Putri, and Setiawan, 2023), and (Kristiyan, Purnomo, and Ropyant 2019), demonstrated that cold pack application effectively minimizes hematoma formation, showing superiority over traditional methods such as sandbag use. While )Valikhani, Mahdizadeh, Eshraghi, Mazloum, and Dehghani, 2020), reported no statistically significant differences between cryotherapy and control groups, their findings may be attributed to shorter application durations. This variation shows how important it is to have a clear and consistent protocol, as highlighted in the randomized controlled trial by ( Sokhanvar, Tirgari, Forouzi, Salari, and Jahani, 2023), which focused on differences in how and when the cold therapy was applied.

Together, these studies highlight the need for continued research to develop standardized, evidence-based protocols for the use of ice bag application in post-PCI care. This study aims to build on existing evidence by evaluating the effectiveness of ice therapy in reducing complications and improving patient outcomes. By doing so, it seeks to promote a simple, practical, and effective method for managing common post-PCI issues-one that can be easily implemented in clinical settings to enhance recovery and increase patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adult patients (aged 18 years and above) who have undergone elective PCI via femoral artery access.

2. Patients who are conscious, oriented, and able to report pain level. 3. Hemodynamically stable post-procedure.

Exclusion Criteria:

* 1. Patients with active infections 2. Patient with double femoral sheath region. 3. Patients with bleeding scar tissue from burns, wounds or hematoma in the femoral artery area before sheath removal.

  4. Patients with known peripheral vascular disease affecting the femoral artery.

  5. Allergy or contraindication to cold application. 6. Active bleeding at the access site. 7. Patients receiving anti-coagulation therapy beyond the standard post-PCI protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain Level | 3 months
  Assessed using a standardized pain scale

SECONDARY OUTCOMES:
Hematoma Formation | 3 months
  Presence and size of hematoma at the puncture site, measured in centimeters using hematoma scale